CLINICAL TRIAL: NCT01969942
Title: A Phase I Study to Examine the Toxicity of Allogeneic Stem Cell Transplantation for Relapsed or Therapy Refractory Ewing Sarcoma
Acronym: ASCT
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: No subjects meeting study inclusion were enrolled.
Sponsor: University of Louisville (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13.0176
Record Dates: First submitted 2013-10-21; First posted 2013-10-25 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Ewing Sarcoma
Keywords: Ewings sarcoma
MeSH Terms: conditions — Sarcoma, Ewing | interventions — fludarabine phosphate; Busulfan; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- allogeneic stem cell transplantation Plan A (Experimental): Subjects will receive the vaccine, Busulfan and Melphalan.
  Interventions: Biological: allogeneic stem cell transplantation; Drug: Busulfan; Drug: Melphalan
- allogeneic stem cell transplantation Plan B (Experimental): If subject have already received a stem cell transplant using Busulfan and Melphalan, they will receive Clysophosohamide and Fludarabine.
  Interventions: Biological: allogeneic stem cell transplantation; Drug: Clyclophosphamide; Drug: Fludarabina

INTERVENTIONS:
Biological: allogeneic stem cell transplantation
Drug: Clyclophosphamide
  Arms: allogeneic stem cell transplantation Plan B
Drug: Fludarabina
  Arms: allogeneic stem cell transplantation Plan B
Drug: Busulfan
  Arms: allogeneic stem cell transplantation Plan A
Drug: Melphalan
  Arms: allogeneic stem cell transplantation Plan A

SUMMARY:
The purpose of this study is to examine the toxicity of using allogeneic stem cell transplantation for treatment of subjects with relapsed or refractory Ewing Sarcoma (ES). Donors will consist of either Human Leukocyte Antigen identical (HLA)or 9/10 (A, B, C, DR, DQ [A, B, C, are Class I markers for HLA and DR and DQ are Class II markers for Matching for Transplant for Donors to match with recipient]) matched related or unrelated donors. Specifically, we will examine:

* The toxicity of allogeneic stem cell transplant (SCT) in this patient population, as related to incidence of grade 3-4 acute Graft Verse Host Disease (GVHD).
* The incidence of transplant related mortality at 100 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 0-30 years with relapsed or therapy refractory Ewings sarcoma, excluding patients with brain metastases. Patients who have received a prior autologous stem cell transplant are eligible.
* Related and unrelated marrow and peripheral blood stem donors must be 9/10 or 10/10 (HLA A, B, C, DR, DQ) matched with the recipient.

Exclusion Criteria:

* Organ dysfunction: Patients who have the following levels of organ system dysfunction are not eligible:

  * Cardiac: Ejection Fraction less than 50 percent
  * Renal: Est. Creatinine Clearance less than 50
  * Hepatic: Bilirubin greater than 3.0
  * Pulmonary: Diffusing Capacity for Carbon Monoxide (DLCO) less than 70 percent, or for patient who cannot cooperate with pulmonary function testing, O2 saturation less than 95 percent on room air.
* Performance status: Lansky performance less than 70; Eastern Cooperative Oncology Group (ECOG) status greater than or equal to 2
* Patients with an isolated recurrence of their tumor (in the site of primary tumor) greater than 1 year after completing therapy are excluded as these patients could be cured with local therapy alone.

  * As part of the standard of care for pre-transplant evaluation subjects will be tested for exposure to viral agents such as hepatitis B, C, HTLV-1/2 and HIV. Subjects testing positive for HI may be rejected as candidates for transplantation, based on the clinical judgement of the stem cell transplant physician.

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2013-04; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Development of Grade 3-4 GVHD | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Lucas, M.D., Principal Investigator — University of Louisville
Locations (1):
- Pediatric Hematology/Oncology University of Louisville, Louisville, Kentucky, United States

REFERENCES:
- See also: University of Louisville Peds--Heme/Onc — https://louisville.edu/medschool/pediatrics/clinical/sections-divisions/hem-onc